CLINICAL TRIAL: NCT03091400
Title: Phase Two Randomized Controlled Crossover Trial of Atomoxetine to Treat Memory Impairment Due to Multiple Sclerosis
Brief Title: Recall Enhancement Through Treatment With Atomoxetine in MS (RETAIN-MS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James F. Sumowski, Assoicate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 16-1552
Record Dates: First submitted 2017-03-16; First posted 2017-03-27 (Actual); Results first posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-02

CONDITIONS: Memory Disorders; Multiple Sclerosis
Keywords: Memory Disorders; Multiple Sclerosis; Atomoxetine Hydrochloride
MeSH Terms: conditions — Memory Disorders; Multiple Sclerosis | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Atomoxetine (Experimental): Atomoxetine (40 mg qd titration dose for first seven days, followed by 80 mg qd target dose for remaining five weeks)
  Interventions: Drug: Atomoxetine
- Placebo (Placebo Comparator): Identically encapsulated placebo, with dose matched to experimental agent (40 mg qd titration dose for first seven days, followed by 80 mg qd target dose for remaining five weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Atomoxetine — Atomoxetine (40 mg qd titration dose for first seven days, followed by 80 mg qd target dose for remaining five weeks)
  Other Names: Strattera (Eli Lilly)
  Arms: Atomoxetine
Drug: Placebo — Identically encapsulated placebo, with dose matched to experimental agent (40 mg qd titration dose for first seven days, followed by 80 mg qd target dose for remaining five weeks)
  Arms: Placebo

SUMMARY:
The purpose of this crossover trial is to investigate whether atomoxetine (versus placebo) improves memory function in persons with memory deficits due to multiple sclerosis.

DETAILED DESCRIPTION:
Approximately half of persons with multiple sclerosis (MS) develop memory decline, which makes it difficult to maintain gainful employment, manage a household, and lead a fully-engaged social life. There are currently no validated symptomatic treatments for memory deficits in persons with MS. The study team will perform a fourteen week double-blind phase-two crossover randomized controlled trial (RCT) of atomoxetine (80mg qd, six weeks) versus placebo (six weeks) to improve memory in MS patients with documented memory impairment (two-week washout between phases). Atomoxetine is a non-stimulant selective norepinephrine reuptake inhibitor FDA-approved to treat cognitive-behavioral symptoms of attention deficit / hyperactivity disorder (ADHD; Strattera, Eli Lilly). Pre-clinical evidence suggests that atomoxetine may also improve memory by targeting brain mechanisms responsible for memory function (norepinephrine in the hippocampus). Twenty-four MS patients demonstrating objective memory impairment on neuropsychological screening tests will be randomly assigned to once-daily orally-administered atomoxetine or identically-encapsulated placebo. After a two-week washout period, patients will be switched to the opposite condition. The RCT will be performed at the Corinne Goldsmith Dickinson Center for MS at the Icahn School of Medicine at Mount Sinai. Baseline and follow-up evaluations will assess change in objective memory function (Primary Outcome), as well as Secondary Outcomes of patient-reported memory change, additional objective measures of memory function, and a measure of speeded symbol-digit coding (the most widely-used test of cognition in persons with MS). Tertiary / Other Outcomes examine sustained attention, processing speed, working memory, fatigue, mood, manual dexterity, and walking speed. The researchers predict that atomoxetine will lead to significantly greater improvements in Primary and Secondary memory outcomes relative to placebo. Consistent with the ADHD literature, there may be additional benefits of atomoxetine versus placebo on measures of attention, processing speed, and working memory. Results of this phase 2 trial will inform decisions / planning for a possible phase 3 trial, which may ultimately support the use of non-stimulant, once-daily atomoxetine as a memory treatment option for MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple Sclerosis based on the Revised McDonald criteria
* Age 21 - 60 years.
* Patient self-report of memory decline from previously higher level of functioning.
* Memory Impairment on validated neuropsychological memory screening tests, as follows:

  1. performance ≤16th percentile on both (i) Rey Auditory Verbal Learning Test (RAVLT) Total Learning (TL) and (ii) WMS-IV Visual Reproduction I (VR-I); and b) mean normative memory performance (RAVLT TL and WMS-IV VR-I) is at least 1.0 standard deviation below expectations based on the Wechsler Test of Adult Reading (WTAR)

Exclusion Criteria:

* Current stimulant medication usage.
* Previous diagnosis or treatment for ADHD or any neurologic condition other than multiple sclerosis (e.g., traumatic brain injury, epilepsy)
* Clinical relapse of MS within 60 days of screening,
* Change in disease-modifying therapy within 90 days of screening,
* Below average estimated premorbid intelligence (WTAR, < 16th percentile),
* Severe cognitive impairment indicated by a Mini-Mental Status Examination (MMSE) < 24/30.
* Contraindications for atomoxetine use: (a) self-reported history of suicidal ideation within the last twelve months (Columbia Suicide Severity Rating Scale), (b) diagnosis of bipolar illness, (c) moderate or severe current depressive symptomatology (Beck Depression Inventory Fast Screen ≥ 9), (d) diagnosis of hepatic disease, (e) narrow angle glaucoma, (f) pheochromocytoma, (g) monoamine oxidase inhibitor within 14 days of study drug start, (h) taking strong CYP2D6 inhibitors (e.g., paroxetine, fluoxetine, quinidine), (i) diagnosis of heart disease, (j) pregnant or planning pregnancy during the study period, (k) breastfeeding, (l) hypersensitivity to atomoxetine or component of formulation.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F Sumowski, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period: 03/16/2017 - 02/20/2018. There was a two-phase screening. Of the 35 participants who met initial screening criteria (e.g., age, MS diagnosis), 24 did not meet secondary screening requirements (e.g., objective memory impairment on assessment). Eleven (11) participants met secondary screening requirements and were randomized.
Groups:
- Atomoxetine Then Placebo: Atomoxetine (40 mg qd titration dose for first seven days, followed by 80 mg qd target dose for remaining five weeks)
  then a two-week washout period, then
  Identically encapsulated placebo, with dose matched to experimental agent (40 mg qd titration dose for first seven days, followed by 80 mg qd target dose for remaining five weeks)
- Placebo Then Atomoxetine: Identically encapsulated placebo, with dose matched to experimental agent (40 mg qd titration dose for first seven days, followed by 80 mg qd target dose for remaining five weeks)
  then a two-week washout period, then
  Atomoxetine (40 mg qd titration dose for first seven days, followed by 80 mg qd target dose for remaining five weeks)
Period: Phase 1 - 6 Weeks
Arm/Group | Atomoxetine Then Placebo | Placebo Then Atomoxetine
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0
Period: Washout - 2 Weeks
Arm/Group | Atomoxetine Then Placebo | Placebo Then Atomoxetine
Started | 5 | 6
Completed | 4 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Phase 2 - 6 Weeks
Arm/Group | Atomoxetine Then Placebo | Placebo Then Atomoxetine
Started | 4 | 6
Completed | 4 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Atomoxetine, Then Placebo: Atomoxetine (40 mg qd titration dose for first seven days, followed by 80 mg qd target dose for remaining five weeks)
  then a two-week washout period, then
  Identically encapsulated placebo, with dose matched to experimental agent (40 mg qd titration dose for first seven days, followed by 80 mg qd target dose for remaining five weeks)
- Placebo, Then Atomoxetine: Identically encapsulated placebo, with dose matched to experimental agent (40 mg qd titration dose for first seven days, followed by 80 mg qd target dose for remaining five weeks)
  then a two-week washout period, then
  Atomoxetine (40 mg qd titration dose for first seven days, followed by 80 mg qd target dose for remaining five weeks)
- Total: Total of all reporting groups
Arm/Group | Atomoxetine, Then Placebo | Placebo, Then Atomoxetine | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (9.1) | 46.0 (5.4) | 44.4 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 1 | 5 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Memory Change
Description: Composite memory function (mean normative z-score) across verbal memory and visuospatial memory tasks: (1) Selective Reminding Test (SRT) assesses verbal learning of a 12-item word list over six trials (a. Total Learning; possible raw score range of 0-72), and recall after a delay (b: Delayed Recall; possible raw score range of 0-36); (2) Brief Visuospatial Memory Test, Revised (BVMT-R; possible raw score range of 0-36) assesses learning of six geometric shapes in six locations over three trials (c. Total Learning), and recall after a delay (d. Delayed Recall; possible raw score range of 0-12). Results reported as composite memory at follow-up minus baseline. Higher scores indicate better outcomes.
Time Frame: baseline and 14 weeks
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 10 | 10
z-score | 0.32 (0.60) | 0.24 (0.46)

2. Secondary Outcome: Change in Patient-Reported Memory Change
Description: Patients will endorse memory change over the past six weeks as: much improved (3), improved (2), slightly improved (1), unchanged (0), slightly worse (-1), worse (-2), much worse (-3).
Time Frame: baseline and 14 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 0.70 (1.16) | 0.90 (1.37)

3. Secondary Outcome: Change in CANTAB Paired Associate Learning
Description: CANTAB Paired Associate Learning (Total Errors Adjusted; possible raw score range of 0-70): a tablet-based memory task requiring subjects to study and recall the location of complex visual images not easily verbalized. Errors are tallied. Results reported as follow-up minus baseline. Higher scores indicate worse outcomes.
Time Frame: baseline and 14 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | -10.30 (11.98) | -8.10 (15.56)

4. Secondary Outcome: Change in NIH Toolbox Picture Sequence Memory Test
Description: NIH Toolbox Picture Sequence Memory Test (possible raw score range of 0-31): a tablet-based task requiring subjects to study the sequence of many activity scenes (e.g., flying a kite) presented visually and audibly. Correct sequences tallied. Results reported as follow-up minus baseline. Higher scores indicate better outcomes.
Time Frame: baseline and 14 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 4.50 (5.80) | 3.20 (2.97)

5. Secondary Outcome: Change in Perceived Deficits Questionnaire (PDQ)
Description: Perceived Deficits Questionnaire (PDQ): the PDQ asks subjects to rate twenty cognitive difficulties on a scale from never (0) to almost always (4). Total ranges from 0-80. Results reported as follow-up minus baseline. Higher scores indicate worse outcomes. If a change is detected, will proceed to identify which of the four subscales were affected: retrospective memory, prospective memory, attention, planning / organization.
Time Frame: baseline and 14 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | -6.60 (9.97) | -5.90 (13.14)

6. Secondary Outcome: Change in Symbol Digit Modalities Test
Description: Symbol Digit Modalities Test (Oral Version, total raw; possible range of 0-110): A test of processing speed requiring subjects to rapidly complete symbol-digit pairings based on a key. Incidental learning may contribute to performance. Total correct in 90 seconds is tallied. Results reported as follow-up minus baseline. Higher scores indicate better outcomes.
Time Frame: baseline and 14 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Atomoxetine | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 7.20 (7.07) | 5.50 (5.42)

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Atomoxetine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 4/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atomoxetine (N=10) | Placebo (N=10)
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Urinary Hesitation (Renal and urinary disorders) | 1 | 0
Pelvic/testicular pain (Reproductive system and breast disorders) | 1 | 0
Painful Urination (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-08): https://cdn.clinicaltrials.gov/large-docs/00/NCT03091400/Prot_SAP_000.pdf